CLINICAL TRIAL: NCT05942586
Title: Systematic Functional Characterization of the Effect of Synbiotic Supplementation with Limosilactobacillus Reuteri PB-W1™ and Prebiotics on Markers of Immune Health, Host Metabolome and Gut Microbiome in Adults with BMI 30-40 Kg/m²
Brief Title: The Symbiont-Restore Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Collaborators: Novozymes A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: APC165
Record Dates: First submitted 2023-06-02; First posted 2023-07-12 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-12

CONDITIONS: Obesity
Keywords: Gut Microbiome; Microbiota; Bacterial Physiological Phenomena; Papua New Guinea; Limosilactobacillus reuteri; Probiotics; Prebiotics; Immunomodulation; Synbiotics; Immune System; Metabolome; Gastrointestinal microbiome; Satiation; Hunger; Dietary fibre; Raffinose; Microbial ecology; Randomised Controlled Trial
MeSH Terms: conditions — Obesity | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: This trial will be conducted as a single-blinded, 2 × 2 factorial design intervention study to systematically compare the effects of the probiotic (L. reuteri PB-W1™), the prebiotic blend (comprising 50 % raffinose and 50 % xylooligosaccharide), the synbiotic (a combination of the probiotic and the prebiotic blend) and relevant placebo controls (maltodextrin in place of the prebiotic blend and placebo capsules in place of the probiotic)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Probiotic Arm (Active Comparator): 30 Participants in this arm will undergo a two-week run-in period consuming placebo sachet (maltodextrin) for the first week and then increasing the dosage in the second week. Following the run-in period, Participants will receive an eight-week intervention consisting of daily consumption of placebo sachets and probiotic capsule containing L. reuteri PB-W1™.
  Interventions: Dietary Supplement: Probiotic capsule (L. reuteri PB-W1™), Placebo sachet
- Prebiotic Arm (Active Comparator): 30 Participants in this arm will undergo a two-week run-in period consuming prebiotic sachets (Prebiotic Blend) for the first week and then increasing the dosage in the second week. During the eight-week intervention, Participants will consume prebiotic sachets three times daily and placebo capsule.
  Interventions: Dietary Supplement: Prebiotic sachet (Prebiotic Blend), Placebo capsule
- Synbiotic Arm (Experimental): 30 Participants in this arm will undergo a two-week run-in period consuming prebiotic sachets (Prebiotic Blend) for the first week and then increasing the dosage in the second week. Following the run-in period, Participants will receive an eight-week intervention consisting of daily consumption of prebiotic sachets, probiotic capsule containing L. reuteri PB-W1™.
  Interventions: Combination Product: Probiotic capsule (L. reuteri PB-W1™), Prebiotic sachet (Prebiotic Blend)
- Placebo Arm (Placebo Comparator): 30 Participants in this arm will undergo a two-week run-in period consuming placebo sachet (maltodextrin) for the first week and then increasing the dosage in the second week. During the eight-week intervention, Participants will consume placebo sachets three times daily and placebo capsule.
  Interventions: Dietary Supplement: Placebo sachet, Placebo capsule

INTERVENTIONS:
Dietary Supplement: Probiotic capsule (L. reuteri PB-W1™), Placebo sachet — Participants in this arm will consume one probiotic capsule (L. reuteri PB-W1™) daily and placebo sachets three times daily (morning, midday, and evening) for a total daily dose of 7.5 g throughout the eight-week intervention period.
  Arms: Probiotic Arm
Dietary Supplement: Prebiotic sachet (Prebiotic Blend), Placebo capsule — Participants in this arm will consume one placebo capsule daily and prebiotic sachets (Prebiotic Blend) three times daily (morning, midday, and evening) for a total daily dose of 15 g throughout the eight-week intervention period.
  Arms: Prebiotic Arm
Combination Product: Probiotic capsule (L. reuteri PB-W1™), Prebiotic sachet (Prebiotic Blend) — Participants in this arm will consume one probiotic capsule (L. reuteri PB-W1™) daily and prebiotic sachets (Prebiotic Blend) three times daily (morning, midday, and evening) for a total daily dose of 15 g throughout the eight-week intervention period.
  Arms: Synbiotic Arm
Dietary Supplement: Placebo sachet, Placebo capsule — Participants in this arm will consume one placebo capsule daily and placebo sachets three times daily (morning, midday, and evening) for a total daily dose of 7.5 g throughout the eight-week intervention period.
  Arms: Placebo Arm

SUMMARY:
Within the framework of the Science Foundation Ireland funded Microbe Restore Project, the Symbiont Restore Study is an Investigator-initiated trial which explores the prospective health advantages associated with a particular bacterium known as Limosilactobacillus reuteri (L. reuteri) PB-W1™.

In the Symbiont Restore Study, we seek to determine if supplementation with L. reuteri PB-W1™, can beneficially alter the composition and function of the gut microbiome, particularly in terms of immunomodulatory benefits, intestinal health, satiety, as well as markers of psychological stress and sleep quality. Additionally, this study will explore whether combining this strain with a prebiotic blend of dietary fibres (comprising 50 % raffinose and 50 % xylooligosaccharide) through a "synbiotic" approach can enhance its therapeutic benefits.

DETAILED DESCRIPTION:
Our preliminary work has shown that the gut microbiome in rural Papua New Guinea (PNG) is more diverse than that of USA controls, and the species Limosilactobacillus reuteri (L. reuteri) was only detectable in PNG. Interestingly, L. reuteri was also regularly detected in humans in studies conducted around 1960, but is very rarely found in contemporary humans, suggesting a recent decline of the L. reuteri population in Westerners. L. reuteri is further convincingly linked to a wide range of health benefits, such as modulating immune function and stimulating immune cell development, and it produces tryptophan metabolites that modulate the immune system.

These findings provide a clear rationale to test the immunological effects of a L. reuteri strain that originates from PNG and explore nutritional strategies to potentially enhance these effects by supporting the colonisation of this strain.

The main objective of this study is to systematically compare the possible immunological effects of synbiotic supplementation with a probiotic, L. reuteri PB-W1™, and a prebiotic blend (comprising 50 % raffinose and 50 % xylooligosaccharide) with that of the probiotic and prebiotic alone and characterise the mechanistic and ecological foundations of any effects.

ELIGIBILITY:
Inclusion Criteria:

* To be considered eligible for enrolment into the study, potential Participants must:

  * Be able to give written informed consent.
  * Be between 18 and 55 years of age.
  * Self-identify as White.
  * Have a BMI of 30-40 kg/m2 and waist circumference of ≥102cm (males) or ≥88cm (females).
  * Have a stable body weight (≤5% change) over the past three months.
  * Be in general good health, as determined by interview and having systolic blood pressure less than 160 mm Hg and diastolic blood pressure less than 100 mm Hg (defined as hypertension stage 2), taken by the investigator.
  * Be willing to avoid consuming dietary supplements, prebiotics, probiotics, or fibre-rich supplements within four weeks prior to the baseline visit and until the end of the study.
  * Be willing to maintain their current level of physical activity.
  * Be willing to consume the investigational product daily for the duration of the study.
  * Be willing to maintain their habitual diet for the duration of the study.

Exclusion Criteria:

* Potential Participants will be excluded from the study if they meet any of the below criteria:

  * Are pregnant, lactating or post-menopausal or women who are planning to become pregnant over the study period.
  * Have hypersensitivity, allergy, or intolerance to any of the components of the investigational products.
  * Have received antibiotic treatment within three months prior to baseline.
  * Are taking a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk, or confound the interpretation of the study results. Participants should have a wash-out period of two-weeks for each of these medications except for antibiotics, which should not have been taken in the previous three months. Participants taking proton pump inhibitors will be allowed into the study if the dose has been stable for at least two months prior to baseline. Similarly, occasional use of over-the-counter non-steroidal analgesics may be acceptable (at the discretion of the Chief Investigator). However, participants will be required to note any medications consumed via the Medical History, Medications and Supplements Log (MR2006).
  * Have a history or indication of drug and/or alcohol abuse at the time of enrolment.
  * Have a significant active and medically diagnosed acute or chronic co-existing illness including metabolic, psychiatric, or gastrointestinal disease (such as diarrhoea, Crohn's disease, ulcerative colitis, IBS, diverticulosis, stomach or duodenal ulcers, hepatitis A/B/C, HIV, cancer etc.). Participants that have a significant family history of such diseases or any other condition which contraindicates, in the investigator's judgement, entry to the study will also be excluded.
  * Habitual consumption of >2 alcoholic beverages/day (>28g ethanol/day).
  * Are vegetarian or vegan, those with a typical fibre intake of >30g/day and those that have used dietary supplements (prebiotics/probiotics) in the month leading up to the study.
  * Have made major dietary changes within three months prior to baseline and those with major lifestyle changes planned during the study (e.g., diet, exercise, extensive travel etc).
  * Those with clinically diagnosed eating disorders.
  * Have active gastrointestinal disorder or previous gastrointestinal surgery.
  * Have a chronic medication treatment (e.g., anti-hypertensive medications) of unstable dosage, defined as having been changed within two months prior to baseline.
  * Are severely immunocompromised (HIV positive, transplant recipients, on any anti-rejection medications, on a systemic-acting steroid for >30 days, or have had chemotherapy or radiotherapy in the last 12 months.
  * Have a malignant disease or any concomitant end-stage organ disease.
  * Have symptomatic illness, that in the opinion of the Investigator, contraindicates entry onto the study.
  * Experienced alarm features such as unexplained weight loss, rectal bleeding, a recent change in bowel habits, or significant abdominal pain within three months prior to baseline.
  * Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial.
  * Participants may not be receiving treatment involving experimental drugs.
  * If the Participant has been in a recent experimental trial, these must have been completed not less than 30 days prior to this study.
  * Any Participant that regularly undertakes rigorous exercise defined by International Physical Activity Questionnaire with a score within category 3, Health Enhancing Physical Activity (HEPA) Active.
  * Individuals with pacemakers or implantable cardioverter defibrillators.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 137 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Immune Profile at 8 Weeks | The assessments will be conducted at baseline (pre-intervention) and at the end of the eight-week intervention period.
  Change from baseline serum cytokine concentrations measured using established methods and immune cell response determined through stimulation assays on peripheral blood mononuclear cells at 8 weeks.

SECONDARY OUTCOMES:
Change from Baseline Faecal Microbiome Composition and Diversity at 8 Weeks | The assessments will be conducted at baseline (pre-intervention) and at the end of the eight-week intervention period.
  Change from baseline gut microbiota composition and diversity at eight weeks, through 16S rRNA gene sequencing of faecal samples.
Change from Baseline Metabolic Profile at 8 Weeks | The assessments will be conducted at baseline (pre-intervention) and at the end of the eight-week intervention period.
  Change from baseline faecal, serum, and urinary metabolite concentrations determined through liquid chromatography-mass spectrometry (LC-MS) at eight weeks.
Change from Baseline Satiety Rating over 8 Week Intervention | Throughout the eight-week intervention period, assessed at specific time points (i.e., weekly) during the study.
  Change from baseline satiety rating over 8 week intervention period, through analysis of Participant responses to the Satiety Labelled Intensity Magnitude (SLIM) scale.
Gastrointestinal Tolerance to Dietary Fibre | Throughout the eight-week intervention period, assessed at specific time points (i.e., weekly) during the study.
  Evaluation of the impact of L. reuteri PB-W1™ supplementation with and without a prebiotic blend on gastrointestinal tolerance to dietary fibres (specifically, the prebiotic blend of 50 % raffinose and 50 % xylooligosaccharide) through monitoring of gastrointestinal symptoms and adverse events.

OTHER OUTCOMES:
Change from Baseline Perceived Stress at 8 Weeks | The assessments will be conducted at baseline (pre-intervention) and at the end of the eight-week intervention period.
  Change from baseline perceived stress levels at 8 weeks, using the Cohen's Perceived Stress Scale (PSS).
Change from Baseline Sleep Quality at 8 Weeks | The assessments will be conducted at baseline (pre-intervention) and at the end of the eight-week intervention period.
  Change from baseline sleep quality at 8 weeks, using a Sleep Quality Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Walter, Principal Investigator — University College Cork
Locations (1):
- University College Cork, Cork, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinez I, Stegen JC, Maldonado-Gomez MX, Eren AM, Siba PM, Greenhill AR, Walter J. The gut microbiota of rural papua new guineans: composition, diversity patterns, and ecological processes. Cell Rep. 2015 Apr 28;11(4):527-38. doi: 10.1016/j.celrep.2015.03.049. Epub 2015 Apr 16. PMID 25892234
- [Background] Walter J, Britton RA, Roos S. Host-microbial symbiosis in the vertebrate gastrointestinal tract and the Lactobacillus reuteri paradigm. Proc Natl Acad Sci U S A. 2011 Mar 15;108 Suppl 1(Suppl 1):4645-52. doi: 10.1073/pnas.1000099107. Epub 2010 Jun 25. PMID 20615995
- [Background] Lorea Baroja M, Kirjavainen PV, Hekmat S, Reid G. Anti-inflammatory effects of probiotic yogurt in inflammatory bowel disease patients. Clin Exp Immunol. 2007 Sep;149(3):470-9. doi: 10.1111/j.1365-2249.2007.03434.x. Epub 2007 Jun 22. PMID 17590176
- [Background] Cervantes-Barragan L, Chai JN, Tianero MD, Di Luccia B, Ahern PP, Merriman J, Cortez VS, Caparon MG, Donia MS, Gilfillan S, Cella M, Gordon JI, Hsieh CS, Colonna M. Lactobacillus reuteri induces gut intraepithelial CD4+CD8alphaalpha+ T cells. Science. 2017 Aug 25;357(6353):806-810. doi: 10.1126/science.aah5825. Epub 2017 Aug 3. PMID 28775213
- [Background] Zelante T, Iannitti RG, Cunha C, De Luca A, Giovannini G, Pieraccini G, Zecchi R, D'Angelo C, Massi-Benedetti C, Fallarino F, Carvalho A, Puccetti P, Romani L. Tryptophan catabolites from microbiota engage aryl hydrocarbon receptor and balance mucosal reactivity via interleukin-22. Immunity. 2013 Aug 22;39(2):372-85. doi: 10.1016/j.immuni.2013.08.003. PMID 23973224
- [Background] Roager HM, Licht TR. Microbial tryptophan catabolites in health and disease. Nat Commun. 2018 Aug 17;9(1):3294. doi: 10.1038/s41467-018-05470-4. PMID 30120222